CLINICAL TRIAL: NCT00504907
Title: A Phase I, Single-Centre, Double-Blind, Placebo-Controlled, Escalating Single Oral Dose, Safety and Tolerability Clinical Trial With BTA9881 in Healthy Subjects
Brief Title: Safety Study of Oral BTA9881 to Treat RSV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biota Scientific Management Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Vaxart (Industry)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTA9881-01
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: RSV
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — BTA9881

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Cohort A (Experimental): Placebo or BTA9881 -10mg
  Interventions: Drug: BTA9881; Drug: Placebo
- Cohort B (Experimental): Placebo or BTA9881 - 10mg
  Interventions: Drug: BTA9881; Drug: Placebo
- Cohort C (Experimental): Placebo or BTA9881 - 25mg
  Interventions: Drug: BTA9881; Drug: Placebo
- Cohort D (Experimental): Placebo or BTA9881 - 50mg
  Interventions: Drug: BTA9881; Drug: Placebo
- Cohort E (Experimental): Placebo or BTA9881 - 100mg
  Interventions: Drug: BTA9881; Drug: Placebo
- Cohort F (Experimental): Placebo or BTA9881 - 200mg
  Interventions: Drug: BTA9881; Drug: Placebo
- Cohort G (Experimental): Placebo or BTA9881 - 400mg
  Interventions: Drug: BTA9881; Drug: Placebo

INTERVENTIONS:
Drug: BTA9881 — Single oral escalating doses
Drug: Placebo

SUMMARY:
This is a placebo-controlled, double-blind, randomised, single dose escalation Phase I clinical trial to determine the safety and tolerability of BTA9881 administered orally to healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects >=18 and <=45 years of age.
2. Individuals who have freely given Informed Consent in writing.
3. Male subjects should use appropriate contraception (e.g. condoms) during the time interval between dosing until three months after dosing. Female subjects must be surgically sterile or post-menopausal (defined as at least two years post cessation of menses and/or follicle-stimulating hormone (FSH) >18 mIU/mL and serum oestradiol <110 pmol/L), or must agree to use two forms of the following contraception: oral contraceptives, or other forms of hormonal birth control including hormonal vaginal rings or transdermal patches, intra-uterine devices, condoms, and spermicide during the time interval between dosing until three months after dosing. Female subjects must also be non-lactating and have a negative serum pregnancy test at screening and at baseline.
4. Able to perform nasal wash procedure.
5. Normotensive (systolic BP ≤ 140 mm Hg and diastolic BP ≤ 90 mm Hg).
6. No abnormal finding of clinical relevance at the screening examination that the Investigator considers might interfere with the objectives of this clinical trial.
7. No clinically relevant abnormality in the ECG; QTc <430 ms (males) or <450 ms (females).
8. Healthy based on medical history, physical examination, 12-lead ECG and clinical laboratory tests, and with no disease that the Investigator regards as clinically relevant.
9. Negative results in Human Immunodeficiency Virus (HIV) antibody, Hepatitis B surface antigen (HBsAg) and Hepatitis C antibody tests.
10. Willingness to abstain from alcohol and caffeine-containing food and beverages for 48 hours prior to dosing and for the duration of the clinical trial.

Exclusion Criteria:

1. Use of any prescription medication (other than allowable oral contraceptives and implanted hormonal contraceptives) during the 14 days prior to dosing.
2. Use of any non-prescription ('over the counter') product, including herbal products, diet aids, hormone supplements, etc., within 14 days prior to dosing.
3. Intake of any investigational drug within 3 months prior to dosing.
4. History or clinical evidence of significant cardiovascular disease (including risk factors for cardiac arrhythmias) or a previous history of any cardiovascular condition that, in the opinion of the investigator, would interfere with the conduct of the trial.
5. History or clinical evidence of significant cerebrovascular, cardiovascular, gastrointestinal, or haematological disease, or myocardial infarction, or a previous history of any other serious underlying disease (including immunocompromised subjects and/or neutropenic subjects) that, in the opinion of the investigator would interfere with the conduct of the clinical trial.
6. History or clinical evidence of significant respiratory disease (including asthma, chronic obstructive pulmonary disease, cystic fibrosis and/or recurrent lower respiratory tract infection), or upper respiratory tract infection within the last month or lower respiratory tract infection within the last three months.
7. History or clinical evidence of renal disease (including renovascular occlusive disease), nephrectomy and/or renal transplant, and/or previous clinically significant laboratory abnormalities of renal function parameters. All subjects with serum creatinine or proteinuria outside the normal laboratory reference range at screening and baseline that are regarded by the Investigator as clinically significant.
8. History or clinical evidence of hepatic disease and/or previous clinically significant laboratory abnormalities of liver function parameters. All subjects with bilirubin, gamma glutamyl transferase (GGT), alanine transaminase (ALT), and aspartate transaminase (AST) outside the normal laboratory reference range at screening and baseline, that are regarded by the Investigator as clinically significant. Subjects known to have experienced elevated liver enzyme values in previous clinical studies will also be excluded.
9. History or clinical evidence of adrenal disease (including Cushing's Syndrome or Addison's disease) or thyroid disease (including hyper or hypothyroidism), and/or previous clinically significant laboratory abnormalities of adrenal or thyroid function parameters. All subjects with thyroid function (TSH, FT4, FT3) outside the normal laboratory reference range at baseline and regarded by the Investigator as clinically significant.
10. Psychiatric or emotional problems that would invalidate the giving of Informed Consent or limit the ability of the subject to comply with clinical trial requirements.
11. Body Mass Index (BMI) ≤18.5 kg/m2 or >=30.0 kg/m2.
12. History of alcohol and/or drug abuse within 1 year prior to screening (verified by drug screening).
13. Receipt of blood or blood products, or loss of 450 mL or more of blood, during the last three months prior to dosing.
14. Unwillingness or inability to provide Informed Consent or to participate satisfactorily for the entire clinical trial period.
15. Subjects who smoke or have been non-smokers for less than 3 months prior to dosing.
16. Subjects who were previously enrolled in this clinical trial.
17. Poor veins, or fear of venipuncture or sight of blood, or known allergy or hypersensitivity to lidocaine.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ascending single oral doses of BTA9881 in healthy adult subjects. | Two weeks

SECONDARY OUTCOMES:
To assess the pharmacokinetics and dose proportionality of BTA9881 after a single oral dose in healthy adult subjects | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hodsman, MD, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia